CLINICAL TRIAL: NCT00978783
Title: Speech Effects of a Speaking Valve Versus External PEEP in Tracheostomized Ventilator-Dependent Neuromuscular Patients
Brief Title: Speech Effects of a Speaking Valve Versus External Positive End-expiratory Pressure (PEEP) in Tracheostomized Ventilator-Dependent Neuromuscular Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Versailles (Other)
Responsible Party: Lofaso Frédéric, MD,PhD, Head of the Physiological Ward, R. Poincaré Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: PMV vs PEEP
Record Dates: First submitted 2009-09-08; First posted 2009-09-17 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Tracheostomy; Mechanical Ventilation
Keywords: Phonation; Tracheostomy; phonation valve; positive end expiratory pressure
MeSH Terms: interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- speaking valve (Active Comparator)
  Interventions: Device: Passy Muir Valve
- Positive end expiratory pressure (Active Comparator)
  Interventions: Device: Positive end expiratory pressure

INTERVENTIONS:
Device: Passy Muir Valve — The Passy Muir Valve was fixed on the tracheostomy tube
  Other Names: phonation valve
  Arms: speaking valve
Device: Positive end expiratory pressure — 5 cm H2O PEEP was adjusted
  Other Names: PEEP
  Arms: Positive end expiratory pressure

SUMMARY:
Background:

Many patients with respiratory failure related to neuromuscular disease receive chronic invasive ventilation through a tracheostomy. Improving quality of life, of which speech is an important component, is a major goal in these patients. The investigators compared the effects on breathing and speech of low-level positive end-expiratory pressure (PEEP, 5 cm H2O) and of a Passy-Muir speaking valve (PMV) during assist-control ventilation.

Methods:

Flow will be measured using a pneumotachograph. Microphone speech recordings were subjected to both quantitative measurements and qualitative assessments; these last consisted of a perceptual score and an intelligibility score determined by two speech therapists using a French adaptation of the Frenchay Dysarthria Assessment.

DETAILED DESCRIPTION:
METHODS

Patients 10 ventilator-dependent patients with neuromuscular disease. All patients will receive mechanical ventilation via a cuffless tracheostomy. The study protocol was approved by our institutional review board, and written informed consent will be obtained from all patients before study inclusion.

Experimental setup Ventilator-delivered flow will be measured using a pneumotachograph (Fleisch #2, Lausanne, Switzerland) and tracheal pressure at the proximal end of the tracheostomy tube using a differential pressure transducer (Validyne MP 45±100 cm H2O, Northridge, CA, USA). To assess patient gas exchange, oxygen saturation (SpO2) will be estimated using pulse oximetry (Ohmeda Biox, BOC Healthcare, Boulder, CO, USA).

Acoustic speech signals will be recorded using three methods. The signals recorded from a microphone (DM202, MDE, Pierron, Sarreguemines, France) positioned 20 cm from the patient's lips were routed to a microcomputer with an AD converter (MP150® and Acqknowledge®, Biopac system, Goleta, CA, USA) that synchronized respiratory data (ventilator flow and tracheal pressure) and acoustic data. The AD converter will digitize respiratory signals at 128 Hz and speech signals at 20 000 Hz. The acoustic signal will be also routed to the Dragon NaturallySpeaking 10® speech recognition system (Nuance; Burlington, MA, USA) with its specific microphone and a laptop computer containing its speech recognition software. Finally, the acoustic signal will be recorded on a digital recorder (DS55, Olympus®, Herodphot, Manage, France) with a signal bandwidth between 50 and 19 000 Hz to allow assessment of fundamental frequency and subsequent qualitative analysis by speech therapists.

Experimental protocol All patients will be receiving ACV, the ventilation mode used in all tracheostomized patients followed at our neuromuscular unit. VI, TI, backup rate, and inspiratory trigger sensitivity will be kept unchanged. Before testing, patients will be familiarized with the use of 5 cm H2O PEEP and of the PMV. These two conditions will be tested in random order. With each condition, the patient first will use the Dragon NaturallySpeaking 10® voice-training menu, which involves reading a text passage for 10 minutes to enable software training. Then, the patient will continuously utter the [a] sound for as long as possible, read a list of words, utter the [a] sound in a glissando from high pitch to low pitch then from low pitch to high pitch, and read a standard text passage.

Data analysis RR, TI, VI, and the volume expired through the tracheostomy tube (VE) will be measured based on the computerized flow signal. The difference between VI and VE will be used as an approximation of the volume expired through the upper airway. Ventilator triggering by the patient will be considered significant when RR exceeded the backup rate by at least 3 cycles/min.

Speech will be evaluated by measuring the mean time spent speaking during the respiratory cycle, time needed to read the text passage, ability of Dragon NaturallySpeaking 10® to accurately recognize the spoken words, and perceptual analyses by two speech therapists blinded to speech condition. The numbers of grammatical and phonological errors made by Dragon NaturallySpeaking 10® during the standard text reading will be compared between PEEP and PMV. The two speech therapists will assess the recordings presented in pairs, with PEEP vs. PMV in random order. The intelligibility scale used will be a French adaptation of the Frenchay Dysarthria Assessment (0 to 8 scale). In addition, the speech therapists will determine a perceptual score on a 0-128 scale developed by the French authors who adapted the Frenchay Dysarthria Assessment.

At the end of each trial, the patients will evaluate subjective respiratory comfort and subjective speech comfort on 10-cm horizontal visual analog scales (VASs).

Statistical analysis All results will be expressed as means±standard deviation (SD). Differences between the two conditions will be assessed using a paired t test. P values <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Neuromuscular patients
* Patients received mechanical ventilation via a cuffless tracheostomy

Exclusion Criteria:

* Acute respiratory failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
text reading duration | 1 hour

SECONDARY OUTCOMES:
respiratory comfort | 1 hour
speech comfort | 2 hours
Dragon NaturallySpeaking 10® system ability to recognise the speech | 30 minutes
Sustained [a] duration | 15 minutes
perceptual score and intelligibility score determined by 2 blinded speech therapists | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Djillali Annane, MD, PhD, Study Chair — CIC-IT, R. Poincaré Hospital
Locations (1):
- Intensive care Ward of R. Poincaré Hospital, Garches, France